CLINICAL TRIAL: NCT03314220
Title: The Effectiveness of Preoperative Preparation for Improving Perioperative Outcomes in Children and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103013
Record Dates: First submitted 2017-10-02; First posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Children Who Underwent Minor Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care plus preoperative preparation (Experimental): experimental group received standard care plus preoperative preparation, which included a tour, a cartoon video depicting a boy's surgical journey and familiarization with medical equipment.
  Interventions: Behavioral: preoperative preparation
- standard care (No Intervention)

INTERVENTIONS:
Behavioral: preoperative preparation — Participants in the experimental group received standard care plus our newly developed, multicomponent family-centered preoperative preparation program. This program included the following: (1) a tour of the preoperative area and recovery room; (2) a 4-min cartoon video entitled 'I am not afraid of surgery,' which was tailored to the child; this video included 29 scenes that depicted a boy's surgical journey with a particular emphasis on strategies for addressing postoperative pain; and (3) familiarization with medical equipment such as name badges, disposable hair caps, anesthetic masks, EKG leads, and pulse oximeters, which were placed on a doll, to help children understand the surgical instruments and promote better cooperation at the time of anesthesia induction.
  Arms: standard care plus preoperative preparation

SUMMARY:
This study aimed to accomplish the following objectives:

1. Develop a family-centered preoperative preparation program.
2. Evaluate the effectiveness of this program in terms of children's preoperative emotional behaviors, postoperative behavior, and posthospital behavior and caregivers' anxiety.

ELIGIBILITY:
Inclusion Criteria:

* aged 3-12 years, received general anesthesia, and admitted for elective outpatient ear, nose and throat, orthopedic, ophthalmology or general surgery.

Exclusion Criteria:

* Children with severe development delay or chronic illness were excluded. Caregivers were excluded if they could not accompany their child to the hospital on the day of the surgery.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2014-05-15 (Actual); Primary Completion 2016-05-15 (Actual); Study Completion 2016-05-15 (Actual)

PRIMARY OUTCOMES:
Children's Emotional Behaviors: The Children's Emotional Manifestation Scale | before the operative day
  to assess children's emotional behaviors during stressful medical situations
Children's Emotional Behaviors: The Children's Emotional Manifestation Scale | the morning in the day of surgery
  to assess children's emotional behaviors during stressful medical situations
Children's Emotional Behaviors: The Children's Emotional Manifestation Scale | at induction of anesthesia
  to assess children's emotional behaviors during stressful medical situations

IPD SHARING:
Plan to Share IPD: No